CLINICAL TRIAL: NCT01070563
Title: Evaluation of Transcranial Doppler Ultrasonography to Guide the Time of Cerebral Angiography for the Brain Death Diagnosis
Brief Title: Transcranial Doppler Ultrasonography and Brain Death
Status: Completed | Type: Observational
Sponsor: Institut d'Anesthesiologie des Alpes Maritimes (Other)
Responsible Party: Orban Jean-Christophe, MD, Nice University Hospital
Other Study IDs: IAAM 2010-1
Record Dates: First submitted 2010-02-12; First posted 2010-02-18 (Estimated); Last update posted 2011-07-04 (Estimated); Status verified 2011-06

CONDITIONS: Brain Dead
Keywords: Brain death; CT angiography; Ultrasonography, doppler, transcranial
MeSH Terms: conditions — Brain Death | interventions — Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Usual: CT angiography is performed 6 hours after the clinical diagnosis of brain death.
- TCD: When the diagnosis of brain death is made, TCD is performed and then every 2 hours until the flow patterns compatible with brain death are found. Then a CT angiography is performed.
  Interventions: Other: Transcranial doppler

INTERVENTIONS:
Other: Transcranial doppler — A TCD is performed on all cerebral arteries (mean cerebral arteries, anterior cerebral arteries, basilar trunk, vertebral arteries and carotid arteries) until a flow pattern compatible with brain death is found
  Groups: TCD

SUMMARY:
In France the diagnosis of brain death relies on electroencephalography (EEG) or cerebral angiography. Concerning the latter a time of 6 hours is mandatory between the clinical diagnosis and the realization of the cerebral computed tomography (CT) angiography. Transcranial doppler (TCD) is not recommended in the french guidelines for the diagnosis of brain death. In other countries, some flow patterns allow to confirm the diagnosis of brain death. The hypothesis of our study is that TCD could shorten the time between the clinical diagnosis of brain death and the realization of the CT angiography.

ELIGIBILITY:
Inclusion Criteria:

* brain death patients

Exclusion Criteria:

* craniectomy
* post anoxia encephalopathy
* no TCD performed before the clinical diagnosis of brain death
* transtemporal approach impossible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients showing brain injury due to stroke or trauma and developping subsequently brain death
Sampling Method: Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2009-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Time between clinical diagnosis of brain death and realization of CT angiography | the outcome is assessed when the CT angiography is performed

SECONDARY OUTCOMES:
Number of CT angiography required for the diagnosis of brain death | the outcome is measured until the diagnosis of brain death is confirmed

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe Orban, MD, Principal Investigator — Nice University Hospital
Locations (1):
- Centre Hospitalier Universitaire de Nice, Nice, France

REFERENCES:
- [Derived] Orban JC, El-Mahjoub A, Rami L, Jambou P, Ichai C. Transcranial Doppler shortens the time between clinical brain death and angiographic confirmation: a randomized trial. Transplantation. 2012 Sep 27;94(6):585-8. doi: 10.1097/TP.0b013e3182612947. PMID 22918218